CLINICAL TRIAL: NCT05434039
Title: Diclofenac Phonophoresis Versus High Power Pain Threshold Ultrasound in Patients With Mechanical Non-specific Neck Pain
Brief Title: Diclofenac Phonophoresis Versus High Power Pain Threshold Ultrasound on Patients With Neck Pain
Acronym: NP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Al Shaymaa Shaaban Abd El Azeim, principle investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: p.t.REC/012/003672
Record Dates: First submitted 2022-06-22; First posted 2022-06-27 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Neck Pain
Keywords: phonophoresis; high power pain threshold ultrasound; neck pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: diclofenac phonophoresis and high power pain threshold
Who Masked: Participant, Outcomes Assessor
Masking Description: random generator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- diclofenac phonophoresis (Experimental): the patients will receive diclofenac phonophoresis and traditional therapy three times a week for four weeks
  Interventions: Other: diclofenac phonophoresis; Other: conventional therapy
- high power pain threshold ultrasound (Experimental): the patients will receive high power pain threshold ultrasound and traditional therapy three times a week for four weeks
  Interventions: Other: high power pain threshold ultrasound; Other: conventional therapy
- conventional therapy (Active Comparator): the patients will receive traditional therapy three times a week for four weeks
  Interventions: Other: conventional therapy

INTERVENTIONS:
Other: diclofenac phonophoresis — the patients will be in comfortable position and apply diclofenac phonophoresis on upper trapezius and suboccipital muscle by ultrasound device. diclofenac gel was applied circularly with a thickness of 2-3 mm. Then ultrasound with was applied with 1 MHz frequency and 1.5 Wt/cm2 power over the trigger points on the trapezius and suboccipital muscle, for 10 min.
  Arms: diclofenac phonophoresis
Other: high power pain threshold ultrasound — the patients will be in comfortable position and The frequency was set to 1 MHz, and the intensity will be increased from 0.5 to 2 until the patient reported an unpleasant sensation. The probe was held there for 4 s; then, the intensity was reduced by 50%, and the probe will be moved over and around the trigger point. This process is done several times for three minutes
  Arms: high power pain threshold ultrasound
Other: conventional therapy — the patient will receive an active range of motion exercise, stretching and strengthening of all cervical muscles

SUMMARY:
the aim of this study is to investigate the effect of diclofenac phonophoresis versus high power pain threshold ultrasound in patients with mechanical non-specific neck pain

DETAILED DESCRIPTION:
Neck pain can be a long-lasting condition, Between half and three quarters of patients with neck pain will experience recurrence within 1-5 years. Costs for the society due to neck pain are consequently high. Neck pain (NP) is one of the common musculoskeletal problems. NP can be caused by the stress over the musculoskeletal system due to postural disorders and may also be associated with other causes such as intervertebral disc herniation, nerve compression, or fracture. Musculoskeletal pain due to trigger points is one of the most prevalent reasons for patients to seek treatment. The aim of physical therapy treatment in patient with myofascial pain syndrome is to reduce the pain and restore normal function. Most physical therapy treatments for MPS are targeted to the deactivation of MTrPs. Physical therapy techniques include manual therapies; such as ischemic compression, spray and stretch, strain and counter strain, muscle energy techniques, trigger point pressure release, transverse friction massage; needling therapies, and other techniques such as thermotherapy, ultrasound therapy , phonophoresis and laser therapy.Due to the semi-solid properties, a special method is needed for transdermal permeation of lidocaine. Therefore, many studies have focused on enhancing the level of transdermal permeation by either changing the physiochemical properties of lidocaine or using physical modalities In particular, there has been considerable interest in transdermal permeation using various methods based on the idea that the amount and depth of transdermal permeation can be increased using various physical modalities. patients with mechanical neck pain will be allocated randomly into three equal groups; group A will receive phonophoresis and traditional therapy, group B will receive high power pain thresholdand traditional therapy and group C will receive traditional therapy

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed as non-specific neck pain with upper trapezius and suboccipital muscles active myofascial trigger points less than 3 months of duration and have these criteria: taut band on palpation, hyper sensible tender spot in the taut band, local twitch response referred pain pattern
2. body mass index from 18 to 25 kg/m2
3. their ages from 18-30

Exclusion Criteria:

1. if they had trigger point injections within the past 6 months
2. history of neck or upper back surgery, trauma or fracture
3. history of a whiplash injury, skin diseases and lesions, any sensory disturbances, any vascular syndromes, neck and back deformities
4. cervical radiculopathy, and diagnosis of fibromyalgia syndrome, skin diseases

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-30 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  The scale that will be used is visual analogue scale ;each subject will be instructed to put point on line from no pain to tolerable pain

SECONDARY OUTCOMES:
cervical range of motion | up to four weeks
  range of cervical will be measured by CROM device
pressure pain threshold | up to four weeks
  pressure pain threshold will be measured by commander algometer
neck disability | up to four weeks
  neck disability will be measured by Arabic neck disability index